CLINICAL TRIAL: NCT02163330
Title: Normal Pressure Hydrocephalus Treatment by Acetazolamide
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty in recruiting participants to the study
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, israel Steiner, Head of Neurology Department, Rabin Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IS 05 - 12
Record Dates: First submitted 2014-04-13; First posted 2014-06-13 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Motor Condition as Measured by Quantified Scale; Cognitive Investigation
MeSH Terms: interventions — Acetazolamide; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Active Comparator): active comparator group will receives 500 mg azetazolamide daily
  Interventions: Drug: Acetazolamide
- sugar pill (Placebo Comparator): placebo comparator group will receives placebo daily.
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Acetazolamide
  Arms: Acetazolamide
Drug: sugar pill
  Arms: sugar pill

SUMMARY:
Normal pressure hydrocephalus (NPH) is an uncommon cause of dementia possibly reversible with treatment. First described in 1965 it consists of a triad of gait disturbance, cognitive deterioration, and urinary incontinence together with enlarged cerebral ventricles and normal cerebrospinal fluid (CSF) pressure. Foregoing trauma and hemorrhage, infection, mass lesions, or aqueductal stenosis can contribute to hydrocephalus. These symptomatic or secondary forms of NPH are not considered here and the focus lies on the idiopathic type (iNPH). Prevalence of iNPH increases significantly with age. General estimates range from 21.9 per 100,000 in total population surveys but increase up to 181.7 per 100,000 for people 70 to 79 years of age. The clinical presentation varies significantly in severity and progression of symptoms. For diagnosis the entire triad does not have to be present. In typical cases gait and balance disturbances appear either before or concurrently with urinary incontinence or the onset of dementia. Current treatment recommendations are based on surgical diversion of CSF , with shunts placed either into the ventricular system or the lumbar subarachnoid space to a distal site, such as the peritoneal or the pleural cavity or the venous system, where the CSF can be reabsorbed . Even though immediate response rate to shunt treatment might be favorable and rates of 80% responders have been reported , the perioperative and long-term morbidity and mortality of CSF shunting procedures are significant. A meta-analysis of 44 articles found that the pooled, mean rate of shunt complication was 38% . Even though acute surgical complication rates are low, shunt dysfunctions and long-term complications are relatively common. Shunt malfunction (20%), subdural hematoma (2-17%), seizure (3-11%), shunt infection (3-6%) and intracerebral hematoma (3%) are the most common complications . In those with good long-term survival, sustained improvement is possible, with a rate of 39% documented after 5 years .In view of the complication rates, the lack of alternative treatment options and clinical studies is surprising. Even though iNPH per definition lacks raised intracranial pressure on spinal tap, monitoring of ICP prior to surgery reveals an increased amount of brief (usually 30 seconds to 1 minute) increases in the static ICP, called Lundberg B waves, in patients which improve by shunt placements . When patients are scheduled for shunt treatment there is a waiting period of several weeks between diagnosis and operation due to congested waiting list.

Acetazolamide (Diamox) has been shown to reduce the production of CSF in clinical cases of raised intracranial pressure . It is considered the drug of choice for the treatment of idiopathic intracranial pressure (pseudotumor cerebri). Intuitively a connection between Acetazolamide as a treatment option in iNPH seems logical. Encouraging case studies have been published previously showing a fascinating improvement and success of treating iNPH with Acetazolamide. A systematic placebo controlled study concerning the use of Acetazolamide in iNPH is missing and would possibly pave the way to an alternative treatment option avoiding surgery and its complications.

ELIGIBILITY:
Inclusion Criteria:

Included will be subjects with a probable diagnosis of iNPH. The diagnosis will be based primarily on presence of gait impairment plus at least one other impairment in urinary symptoms, cognition impairment or both.

1. Are 60 years old or older
2. Patients who understand the study protocol
3. Patients who meet the criteria for NPH

   1. A typical personal history
   2. A typical brain imaging on head CT or MRI
   3. Normal LP findings excluding other conditions
   4. Exclusion of other conditions causing the symptomatology
   5. Patients who underwent Continuous lumbar drainage or spinal tap which improved symptomatology.

Exclusion Criteria:

1. Patients below the age of 60 years.
2. Patients who underwent shunt surgery
3. Patients with a concurrent diagnosis of a neurodegenerative or neurovascular disease that causes a significant impairment of gait and cognitive functions
4. Patients with symptom duration of more than 6 month
5. Patients with contraindications for acetazolamide treatment:

   * Cirrhosis or marked liver disease or dysfunction
   * hyperchloremic acidosis
   * hypersensitivity to acetazolamide or any component of the product
   * hypersensitivity to sulfonamides or other sulfonamide derivatives, as cross-sensitivity may occur
   * hypokalemia
   * hyponatremia
   * renal dysfunction or disease
   * suprarenal gland failure

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
1. Changes from baseline in motor on the Boon scale at week 4 | Baseline, Week4
  The effect of acetazolamide on motor and cognitive function in iNPH patients will be examined.
  Motor system investigations - Gait assessment using a quantified scale (Boon et al., 1997). Scores from this metric represent 3 summed subscores: 10-m step count, 10-m time, and the following 10 features: hesitation, wide and small steps, low clearance, impaired turning, sway, fall tendency, impaired tandem walking, and inability to walk with and without assistance. The summed score has a range from 2-40, with 2 representing unimpaired gait.

SECONDARY OUTCOMES:
Changes from baseline in cognitive function on the Mattis Dementia Rating Scale (MDRS) and the Montreal Cognitive Assessment (MoCA) | Baseline, week4
  Cognitive tests -Mattis Dementia Rating Scale (MDRS) and Montreal Cognitive Assessment (MoCA) will be performed by our neuropsychology staff.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petach Tiqva, Central District, Israel